CLINICAL TRIAL: NCT06123442
Title: Feasibility and Acceptability of Cognitive Resilience Intervention as a Recovery Therapy for Mental Health Among University Students: A Study Protocol for a Randomized Controlled Clinical Trial
Brief Title: Cognitive Resilience Intervention as a Recovery Therapy for Mental Health
Acronym: CRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2023-1-63
Record Dates: First submitted 2023-10-25; First posted 2023-11-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Reduction in Mental Health and Suicide Are the Focus of Interest; Four Assessment Time Points Would be Used to Monitor Participants Through a Laid Down Conditions
Keywords: "Anxiety"; "Cognitive Resilience"; "Depression"; "Intervention Development"; "suicidal Ideations"; "Students"
MeSH Terms: conditions — Anxiety Disorders; Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: This open-label, 2-year pilot study seeks to determine the feasibility and acceptability of CRI in students with psychological distress comorbid with suicide behavior. This study will employ three single-arm trials followed by a pilot randomized controlled trial with an experimental and control group. This university-based research will use a pretest-posttest design to collect data
Masking Description: After enrolling participants and conducting baseline assessments, individuals will be randomly assigned to one of two treatment conditions using a 1:1 allocation ratio following the guidelines already laid down guidelines. It's worth noting that this study will involve university students from various levels and programs, as long as they meet the criteria outlined in Table 1.2. While the facilitators will be aware of the treatment conditions, the research assistant responsible for conducting assessments after randomization will remain blind to these conditions. The process of characterizing the participants will follow the same approach as the three one-arm trials, with any necessary adjustments made based on lessons learned during the trial groups' execution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- three one-arm trials (N = 4-6/trial) (Experimental): This research protocol entails three one-arm trials and a pilot RCT with 58 participants. Its primary aim is to develop the Cognitive Resilience Intervention (CRI) and assess its feasibility and acceptability. Student feedback and data on feasibility and acceptability will be collected before and after each trial to fine-tune the intervention using empirical guidance. CRI aims to help participants lead more meaningful lives, emphasizing purpose, autonomy, and the pursuit of goals while avoiding suicidal ideation. In contrast, the comparator RCT's control group will undergo General Psychoeducation (GPE), a structured program focusing on enhancing mental health awareness through psychology psycho-education sessions.
  Interventions: Behavioral: Cognitive Resilience Intervention

INTERVENTIONS:
Behavioral: Cognitive Resilience Intervention — Participants will have 12 weeks to complete the program, and then before the post-assessment, there will be a one-month feedback period [22]. This includes twelve components: 1) preliminary routine, 2) significance of knowing yourself, 3) interpreting events and stressors, 4) taking autonomy over events, 5) practicing mindfulness and self-compassion, 6) learning adaptation skills, 7) building connection , 8) purpose in life and personal growth, 9) Regulation and disclosure of emotions, 10) practicing gratitude, and 11) positive Communication both intra and interpersonal, 12) overcoming obstacles and moving forward (in the context of current problems) and the conclusion/retrospection are addressed in 12 sessions while closure and post assessment will be done after a month
  Other Names: CRI

SUMMARY:
The goal of this randomized controlled trial (RCT) is to develop and test a cognitive resilience intervention (CRI) among selected students who are having problems with anxiety, depression, and suicidal thoughts (psychological distress comorbid with suicidal episodes [PDSE]) and to see if it can help lower PDSE among the students who were enrolled. This study will assess the feasibility and acceptability of a CRI among students dealing with anxiety, depression, and suicidal thoughts (psychological distress comorbid with suicidal episodes [PDSE]) and determine if it is effective at reducing PDSE among the sampled students using psychological assessment tools. Participants will be exposed to CRI in the experimental group and psychoeducation in the control group. Researchers will compare the experimental group with the control group and infer the difference between these groups both at the pretest and posttest phases, as well as ascertain the feasibility and acceptability of this therapy among selected participants.

DETAILED DESCRIPTION:
In a bid to assess the feasibility and acceptability of Cognitive Resilience Intervention (CRI) in students with Persistent Distressing Suicidal Ideation (PDSE), this two-year pilot study is designed as an open-label exploration. The study comprises three individual trials, each involving a single group, followed by a pilot randomized controlled trial (RCT) with both experimental and control groups. This research, carried out at the University Psychological Care Services (SUAPSI) of the Autonomous University of Ciudad Juárez, Chihuahua, Mexico, aims to gather data utilizing a pretest-posttest approach.

Participants for the trials and pilot RCT will be recruited through advertisements on the UACJ and SUAPSI websites, as well as through the distribution of flyers. To ensure eligibility, pre-screening and verification of institutional affiliation will be conducted. All participants will be required to provide informed consent before their participation. Clinical assessments, including the Plutchik Suicide Risk Scale (PSRS), General Anxiety Disorder-2 (GAD-2), Patient Health Questionnaire-2 (PHQ-2), and the Brief Resilience Scale (BRS), will be utilized to evaluate participants' eligibility and characteristics. If potential participants do not respond after pre-screening, multiple contact attempts will be made before their participation is terminated.

To ensure equitable distribution of participants across age and gender categories, a restricted randomization method will be employed, dividing participants into three cohorts. A total of 19 participants will be evenly divided between the two groups using randomized block calculations. This approach is aimed at mitigating potential attrition risks and ensuring the desired sample size for the CRI one-arm trials. It is a commonly used method in small RCTs to maintain unbiased selection and comparability between control and treatment groups.

The inclusion and exclusion criteria for the one-arm trials and pilot RCT are the same, although the criteria for the pilot RCT may be adjusted based on lessons learned from the one-arm trials. The primary outcome measures of this study are focused on assessing personal recovery from suicidal ideation and risk factors, with four assessment time points throughout the one-year PDSE period. The Plutchik Suicide Risk Scale (PSRS) and Brief Resilience Scale (BRS) are used to evaluate these outcomes.

Additionally, secondary outcome measures include the General Anxiety Disorder-2 (GAD-2), which assesses core anxiety symptoms. The CRI group, consisting of 19 participants, will meet weekly over 12 weeks, facilitated by the researcher and co-doctorate student colleagues. Qualitative data will be collected from participants and facilitators after each session.

A pilot RCT will be conducted using treatment materials refined through the one-arm trials. Participants and SUAPSI authority will be informed of the readiness for the pilot RCT. Participants will be recruited following the guidelines mentioned in Section 2.2.

In the pilot RCT, participants will be randomly assigned to treatment conditions, while the research assistant conducting assessments will remain blind to these conditions. This study encompasses university students from various levels and programs who meet the criteria outlined in Table 1.2. The process for characterizing participants will mirror the approach used in the one-arm trials, with adjustments based on lessons learned during their execution.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* He or she is current students of UACJ and residence in the Juárez city
* As determined by the mental health treatment provider, sufficient clinical stability and suitability for group therapy.
* Adequate medical stability as determined by a medical professional.
* Imminent history or risk of mental health and suicidal (that is, suicide attempt) or homicidal behavior.
* Suicidal episode within the past weeks (determined by the PSRS inclusion criteria items).
* Scoring 1 above the cut off scores of PSRS, GAD-2, PHQ-2 and scoring low on the BRS

Exclusion Criteria:

* Inability to perform CRI tasks based on their performance on a sample reading and writing task from the manual (given during screening)
* Non-Spanish speaking students
* Lack of capacity to consent or sign the informed consent
* Unable to attend outpatient group treatment program
* Participation in another CRI intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All gender identities are eligible.
Enrollment: 100 (Estimated)
Dates: Start 2024-02-13 (Estimated); Primary Completion 2024-08-13 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The Plutchik Suicide Risk Scale for suicidal risk | 5minutes
  The Plutchik Suicide Risk Scale to measure suicidal ideation; a score of 6 or more indicate the presence of suicidal risk
Brief Resilience Scale for assessing resilient behavior | 1 minute
  The Brief Resilience Scale measures resilience; the scale is a five-point Likert scale ranging from strongly disagree (1) to strongly agree (5). The addition of value (1-5) responses for the 6-item scale range from 6-30. For the final score, responses are divided by the total number of questions answered. Scores are interpreted as follows: Low resilience (1.00-2.99), Normal resilience (3.00-4.30), and High resilience (4.31-5.00). High scores indicate resilience.

SECONDARY OUTCOMES:
The General Anxiety Disorder-2 is for measuring general anxiety | 1 minute
  The General Anxiety Disorder-2 is scored by assigning 0, 1, 2, and 3 for each response category and adding them together. The score ranges from 0 to 6, and scores of 0-2 indicate mild anxiety, but scores of 3 and above indicate generalized anxiety disorder symptoms.
The Patient Health Questionnaire for depression | 1 minute
  The Patient Health Questionnaire for measuring depression is scored by assigning 0, 1, 2, and 3 for each response category and adding them together. The score ranges from 0 to 6, and scores of 0-2 indicate mild depression; a score of 3 or greater is considered positive for depression

OTHER OUTCOMES:
Client Satisfaction Questionnaire for assessing the satisfaction on therapy received | 4minutes
  The Client Satisfaction Questionnaire has a 4-point response range from "1" for low satisfaction to "4" for high satisfaction. The scale scores range from 0 to 32 points; a score of 6 or greater is suggestive of client satisfaction with therapy outcomes; higher scores indicate greater satisfaction.
The Competence Scale for Psychoeducation for Facilitator Competency | 4 minutes
  The Competence Scale for Psychoeducation used a 7-point rating scale (0=poor, 1=barely adequate, 2=mediocre, 3=satisfactory, 4=good, 5=very good, and 6=excellent). The score for therapists' competence is 31 and above; a higher score indicates a greater level of competence.

CONTACTS AND LOCATIONS:
Overall Officials: Rotimi Oguntayo, Mphil, Principal Investigator — Universidad Autonoma de Ciudad Juarez; Verónica Portillo-Reyes, PhD, Study Chair — Universidad Autonoma de Ciudad Juarez; Gerardo Ochoa Meza, PhD, Study Chair — Universidad Autonoma de Ciudad Juarez; Marisela Gutiérrez-Vega, PhD, Study Director — Universidad Autonoma de Ciudad Juarez
Locations (1):
- SUAPSI, Juárez, Chihuahua, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The study will make available the procedure for collecting data at the pre-test, intervention, and post-test levels.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2023-2024
Access Criteria: The manuscript and the published copy will be made available upon reasonable request.